CLINICAL TRIAL: NCT03898180
Title: A Phase 3, Randomized, Double-blind Study to Compare the Efficacy and Safety of Pembrolizumab (MK-3475) in Combination With Lenvatinib (E7080/MK-7902) Versus Pembrolizumab and Placebo as First Line Treatment for Locally Advanced or Metastatic Urothelial Carcinoma in Cisplatin-ineligible Participants Whose Tumors Express PD-L1, and in Participants Ineligible for Any Platinum-containing Chemotherapy Regardless of PD-L1 Expression (LEAP-011)
Brief Title: Study of First-line Pembrolizumab (MK-3475) With Lenvatinib (MK-7902/E7080) in Urothelial Carcinoma Cisplatin-ineligible Participants Whose Tumors Express Programmed Cell Death-Ligand 1 and in Participants Ineligible for Platinum-containing Chemotherapy (MK-7902-011/E7080-G000-317/ LEAP-011)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7902-011; MK-7902-011 (Other: Merck); E7080-G000-317 (Other: Eisai); LEAP-011 (Other: Merck); 194808 (Registry Identifier: JAPIC-CTI); 2018-003752-21 (EudraCT Number)
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Results first posted 2023-10-31 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Urothelial Carcinoma
Keywords: Advanced or metastatic urothelial cancer; Lenvatinib; Pembrolizumab; Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Transitional Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study was unblinded with Amendment 3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Lenvatinib (Experimental): Participants receive pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to ~2 years) PLUS lenvatinib 20 mg via oral capsule once daily (QD) until progressive disease or discontinuation. With protocol amendment 3 (effective: Sep-24-2021), participants discontinue lenvatinib.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib
- Pembrolizumab + Placebo (Active Comparator): Participants receive pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to ~2 years) PLUS placebo for lenvatinib via oral capsule QD until progressive disease or discontinuation. With protocol amendment 3 (effective: Sep-24-2021), participants discontinue placebo.
  Interventions: Biological: Pembrolizumab; Drug: Placebo for lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
Drug: Lenvatinib — oral capsule
  Other Names: MK-7902; E7080; LENVIMA®
  Arms: Pembrolizumab + Lenvatinib
Drug: Placebo for lenvatinib — oral capsule
  Arms: Pembrolizumab + Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of lenvatinib (MK-7902/E7080) in combination with pembrolizumab (MK-3475) in the treatment of cisplatin-ineligible participants with a Programmed Cell Death-Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥10, or in participants ineligible for any platinum-containing chemotherapy regardless of CPS, with advanced/unresectable or metastatic urothelial carcinoma (UC).

The primary hypotheses for this study are that:

1. Pembrolizumab + lenvatinib is superior to pembrolizumab + placebo with respect to Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by blinded independent central review (BICR), and
2. Pembrolizumab + lenvatinib is superior to pembrolizumab + placebo with respect to Overall Survival (OS).

Based on recommendation of the external Data Monitoring Committee (eDMC), Amendment 3 (effective: September [Sep]-24-2021) was implemented to unblind the study and discontinue lenvatinib and placebo treatment. The eDMC was then disbanded.

With Amendment 4 (effective: December-5-2022) second course pembrolizumab will no longer be offered. Any participant receiving second course pembrolizumab treatment prior to initiation of Amendment 4 will be able to complete treatment as planned. Study participation will end after the final administration of pembrolizumab. Participants who either complete 35 administrations of pembrolizumab or discontinue pembrolizumab will discontinue from the study following the safety follow-up visit. AEs and spontaneously reported pregnancies will be reported and followed per protocol. The overall study ends when the last participant completes the last study-related contact or visit, withdraws from the study, or is lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of advanced/unresectable (inoperable) or metastatic urothelial carcinoma (UC) of the renal pelvis, ureter (upper urinary tract), bladder, or urethra.
* Has ≥1 measurable target lesion per RECIST 1.1 as assessed by the local site investigator/radiologist.
* Has provided an archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated and adequate for Programmed Death-Ligand 1 (PD-L1) evaluation.
* Has received no prior systemic chemotherapy for advanced or metastatic UC with the following exceptions:
* Neoadjuvant (prior to surgery) platinum-based chemotherapy for treatment of muscle-invasive bladder cancer with recurrence >12 months from completion of the therapy is permitted.
* Adjuvant (following surgery) platinum-based chemotherapy following radical cystectomy, with recurrence >12 months from completion of the therapy, is permitted.
* Meets criteria for either option a or option b (below):
* a. Has a tumor(s) with PD-L1 combined positive score (CPS) ≥10 and is considered ineligible to receive cisplatin-based combination therapy, based on 1 of the following:
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 2 within 7 days prior to randomization
* National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 Grade ≥2 audiometric hearing loss
* NCI CTCAE Version 4.0 Grade ≥2 peripheral neuropathy OR
* b. In the opinion of the investigator, is considered ineligible to receive any platinum-based chemotherapy (i.e., ineligible for cisplatin and carboplatin) based on:
* ECOG PS of 2 within 7 days prior to randomization and ≥1 of the following:
* Documented visceral metastatic disease
* NCI CTCAE Version 4.0 Grade ≥2 audiometric hearing loss
* NCI CTCAE Version 4.0 Grade ≥2 peripheral neuropathy
* Other reason for the participant's being unable to receive both cisplatin and carboplatin safely. Additional criteria for platinum ineligibility will be considered and allowed on a case-by-case basis, following consultation with the Sponsor. Note: Participants considered ineligible for any platinum-based chemotherapy are eligible for this study regardless of their tumor PD-L1 status.
* Has ECOG PS 0, 1, or 2 within 7 days prior to randomization and a life expectancy of ≥3 months.
* Male participants are eligible to participate if they agree to the following during the treatment period and for ≥30 days after the last dose of pembrolizumab or lenvatinib/placebo:
* Be abstinent from heterosexual intercourse as their preferred and usual lifestyle and agree to remain abstinent, OR
* Must agree to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause as detailed below:
* Agrees to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant. Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile-vaginal penetration.
* A female participant is eligible to participate if she is not pregnant or breastfeeding and if she is not a WOCBP OR is a WOCBP and is using a contraceptive method that is highly effective (with a failure rate of <1% per year) with low user dependency, or is abstinent from heterosexual intercourse as her preferred and usual lifestyle during the intervention period and for ≥120 days post pembrolizumab or ≥30 days post lenvatinib/placebo.
* Has adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mm Hg at screening and no change in antihypertensive medications within 1 week prior to randomization.
* Has adequate organ function.

Exclusion Criteria:

* Has disease that is suitable for local therapy administered with curative intent (e.g. chemotherapy and radiation for Stage 3 disease).
* Has tumor with any neuroendocrine or small cell component.
* Has a history of a gastrointestinal condition or procedure (e.g. gastric bypass, malabsorption) that, in the opinion of the investigator, may affect oral drug absorption.
* Has had major surgery within 3 weeks prior to the first dose of study treatment
* Has a pre-existing Grade ≥3 gastrointestinal or non-gastrointestinal fistula.
* Has radiographic evidence of major blood vessel invasion/infiltration, or has had clinically significant hemoptysis (≥0.5 teaspoon of bright red blood) or tumor bleeding within 2 weeks prior to the first dose of study treatment.
* Has had significant cardiovascular impairment within 12 months of the first dose of study treatment, such as history of New York Heart Association (NYHA) >Class II congestive heart failure, unstable angina, myocardial infarction or cerebrovascular accident (CVA)/stroke, cardiac revascularization procedure, or cardiac arrhythmia associated with hemodynamic instability.
* Has known intolerance or severe hypersensitivity (Grade ≥3) to pembrolizumab or lenvatinib or any of their excipients
* Has received lenvatinib as monotherapy or in combination with a programmed cell death-1/programmed cell death-ligand 1 (PD-1/PD-L1) inhibitor or has previously been enrolled in a clinical study evaluating lenvatinib for bladder cancer, regardless of the treatment received.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 inhibitor, indoleamine-pyrrole 2,3 dioxygenase (IDO1) inhibitor, or agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated antigen 4 [CTLA-4], OX 40, CD137), or any other antibody or drug targeting T-cell costimulatory pathways in the adjuvant or advanced/metastatic setting.
* Has received prior radiotherapy to a metastatic site without the use of chemotherapy radiosensitization within 3 weeks of the first dose of study treatment, with the exception of palliative radiotherapy to bone lesions, which is allowed if completed 2 weeks before the start of study treatment. Participants must have recovered from all radiation-related toxicities, and must not require corticosteroids.
* Has received a live vaccine within 30 days prior to the first dose of study treatment.
* In the investigator's judgment, has not recovered from toxicity or other complications from any major surgery prior to starting study treatment.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Has history or presence of an abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (at a dose exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to randomization.
* Has had an active malignancy (except locally advanced or metastatic UC) within the past 36 months. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) who have undergone potentially curative therapy are not excluded.
* Has a history of prostate cancer (T2NXMX or lower with Gleason score ≤7) treated with definitive intent (surgically or with radiation therapy) ≥1 year prior to study entry is acceptable, provided that the participant is considered prostate cancer-free.
* Has central nervous system (CNS) metastases, unless the participant has completed local therapy (e.g. whole brain radiation therapy, surgery, or radiosurgery) and has discontinued use of corticosteroids for this indication for ≥4 weeks before starting study treatment. Any signs (e.g. radiologic) or symptoms of CNS metastases must be stable for ≥4 weeks before starting study treatment.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with disease-modifying agents, corticosteroids, or immunosuppressive drugs).
* Has a history of (non-infectious) pneumonitis that required systemic steroids, or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of or is positive for active hepatitis B virus (HBV) or has active hepatitis C virus (HCV).
* Has active tuberculosis (TB).
* Is receiving hemodialysis.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of pembrolizumab and lenvatinib/placebo.
* Has had an allogeneic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (194):
- United States (21):
  - Banner MD Anderson Cancer Center ( Site 0016), Gilbert, Arizona
  - Community Cancer Institute ( Site 0777), Clovis, California
  - University of California Irvine Medical Center ( Site 0078), Orange, California
  - John Wayne Cancer Institute ( Site 0017), Santa Monica, California
  - Northwest Georgia Oncology Centers PC ( Site 0707), Marietta, Georgia
  - University of Chicago ( Site 0039), Chicago, Illinois
  - Joliet Oncology Hematology ( Site 0091), Joliet, Illinois
  - Quincy Medical Group ( Site 0022), Quincy, Illinois
  - New England Cancer Specialists ( Site 0047), Scarborough, Maine
  - Karmanos Cancer Institute ( Site 0712), Detroit, Michigan
  - Mercy Hospital Saint Louis - David C. Pratt Cancer Center ( Site 0095), St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada ( Site 0005), Las Vegas, Nevada
  - St. Peter's Hospital Cancer Care Center ( Site 0042), Albany, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health ( Site 0002), New York, New York
  - Oklahoma Cancer Specialists and Research Institute, LLC ( Site 0774), Tulsa, Oklahoma
  - Thomas Jefferson University Hospital ( Site 0051), Philadelphia, Pennsylvania
  - Medical University of South Carolina-Hollings Cancer Center ( Site 0029), Charleston, South Carolina
  - Baylor Scott & White Medical Center - Temple ( Site 0706), Temple, Texas
  - Virginia Cancer Institute ( Site 0099), Richmond, Virginia
  - Seattle Cancer Care Alliance ( Site 0003), Seattle, Washington
  - Cancer Care Northwest ( Site 0009), Spokane, Washington
- Argentina (9):
  - Centro de Oncologia e Investigacion Buenos Aires COIBA ( Site 0577), Berazategui, Buenos Aires
  - Centro de Urología CDU ( Site 0590), Buenos Aires, Buenos Aires F.D.
  - Instituto Medico Alexander Fleming ( Site 0578), Buenos Aires, Buenos Aires F.D.
  - Centro de Investigaciones Clinicas - Clinica Viedma ( Site 0585), Viedma, Río Negro Province
  - Centro Oncológico de Rosario ( Site 0584), Rosario, Santa Fe Province
  - Instituto de Investigaciones Metabolicas ( Site 0589), Buenos Aires
  - Centro Medico Dra De Salvo ( Site 0593), Buenos Aires
  - CEMAIC ( Site 0581), Córdoba
  - Centro Oncologico de Integracion Regional. COIR ( Site 0576), Mendoza
- Australia (5):
  - Macquarie University ( Site 0151), North Ryde, New South Wales
  - Mater Misericordiae Ltd ( Site 0158), South Brisbane, Queensland
  - Monash Health ( Site 0160), Clayton, Victoria
  - Peninsula Health Frankston Hospital ( Site 0153), Frankston, Victoria
  - Austin Health-Austin Hospital ( Site 0154), Heidelberg, Victoria
- Canada (5):
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0101), Hamilton, Ontario
  - Lakeridge Health ( Site 0103), Oshawa, Ontario
  - Sunnybrook Research Institute ( Site 0106), Toronto, Ontario
  - CHUQ-Univ Laval-Hotel Dieu de Quebec ( Site 0104), Québec, Quebec
  - CIUSSS de l Estrie Centre Hospitalier Universitaire de Sherbrooke ( Site 0102), Sherbrooke, Quebec
- China (18):
  - Peking University First Hospital ( Site 0726), Beijing, Beijing Municipality
  - Fifth Medical Center of CPLA General Hospital ( Site 0732), Beijing, Beijing Municipality
  - Peking University Third Hospital ( Site 0727), Beijing, Beijing Municipality
  - Chongqing Cancer Hospital ( Site 0741), Chongging, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University ( Site 0743), Xiamen, Fujian
  - Sun Yat-Sen University Cancer Center ( Site 0752), Guangdong, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University ( Site 0749), Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University ( Site 0746), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital ( Site 0750), Harbin, Heilongjiang
  - Hubei Cancer Hospital ( Site 0744), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 0745), Changsha, Hunan
  - Nanjing Drum Tower Hospital ( Site 0737), Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center ( Site 0721), Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University ( Site 0725), Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 0738), Xian, Shanxi
  - Cancer Hospital Affiliated to Xinjiang Medical University ( Site 0751), Ürümqi, Xinjiang
  - Second Affiliated Hospital, Zhejiang University ( Site 0734), Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital ( Site 0735), Hangzhou, Zhejiang
- Denmark (5):
  - Rigshospitalet ( Site 0680), Copenhagen, Capital Region
  - Herlev Hospital ( Site 0681), Herlev, Capital Region
  - Aarhus Universitets hospital ( Site 0683), Aarhus N, Central Jutland
  - Aalborg Universitets Hospital ( Site 0684), Aalborg, North Denmark
  - Odense Universitetshospital ( Site 0682), Odense, Region Syddanmark
- France (15):
  - CHU Poitiers ( Site 0253), Poitiers, Ain
  - Institut de Cancerologie Strasbourg Europe ( Site 0232), Strasbourg, Alsace
  - Hopital de la Timone ( Site 0246), Marseille, Bouches-du-Rhone
  - CHIC Quimper ( Site 0245), Quimper, Finistere
  - CHU de Bordeaux- Hopital Saint Andre ( Site 0235), Bordeaux, Gironde
  - Clinique Pasteur ( Site 0252), Tolouse, Haute-Garonne
  - Centre de Cancerologie du Grand Montpellier ( Site 0249), Montpellier, Languedoc-Roussillon
  - Centre Rene Gauducheau ICO ( Site 0250), Saint-Herblain, Loire-Atlantique
  - Institut de Cancerologie de l Ouest Site Paul Papin ( Site 0236), Angers, Maine-et-Loire
  - Centre D Oncologie de Gentilly ( Site 0240), Nancy, Meurthe-et-Moselle
  - Centre Hospitalier de la Cote Basque ( Site 0239), Bayonne, Pyrenees-Atlantiques
  - Centre Leon Berard ( Site 0244), Lyon, Rhone
  - Institut Gustave Roussy ( Site 0243), Villejuif, Val-de-Marne
  - CHD Vendee-onco-hematologie ( Site 0251), La Roche-sur-Yon, Vendee
  - Institut Curie ( Site 0237), Paris
- Germany (8):
  - Klinikum der Eberhard-Karls-Universitaet Tuebingen ( Site 0271), Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Giessen und Marburg GmbH ( Site 0284), Marburg, Hesse
  - Universitaetsmedizin Goettingen ( Site 0281), Göttingen, Lower Saxony
  - Helios Kliniken Schwerin GmbH ( Site 0278), Schwerin, Mecklenburg-Vorpommern
  - Universitaetsklinikum Essen ( Site 0274), Essen, North Rhine-Westphalia
  - Staedtisches Krankenhaus Kiel GmbH ( Site 0285), Kiel, Schleswig-Holstein
  - Universitaetsklinikum Schleswig-Holstein-Campus Lubeck ( Site 0277), Lübeck, Schleswig-Holstein
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 0282), Hamburg
- Hungary (8):
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Okta-Klinikai Onkológiai és Sugárterápiás Ce, Miskolc, Borsod-Abauj Zemplen county
  - Bacs-Kiskun Megyei Korhaz ( Site 0510), Kecskemét, Bács-Kiskun county
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet ( Site 0507), Szolnok, Jász-Nagykun-Szolnok
  - Markusovszky Egyetemi Oktatokorhaz ( Site 0502), Szombathely, Vas County
  - Bajcsy Zsilinszki Korhaz es Rendelointezet ( Site 0509), Budapest
  - Orszagos Onkologiai Intezet ( Site 0503), Budapest
  - Uzsoki Utcai Korhaz ( Site 0508), Budapest
  - Somogy Megyei Kaposi Mor Oktato Korhaz ( Site 0504), Kaposvár
- Israel (10):
  - Ha Emek Medical Center ( Site 0560), Afula
  - Assuta Ashdod Public ( Site 0562), Ashdod
  - Rambam Medical Center ( Site 0552), Haifa
  - Shaare Zedek Medical Center ( Site 0559), Jerusalem
  - Hadassah Ein Kerem Medical Center ( Site 0558), Jerusalem
  - Meir Medical Center ( Site 0554), Kfar Saba
  - Rabin Medical Center ( Site 0553), Petah Tikva
  - Sheba Medical Center ( Site 0551), Ramat Gan
  - Sourasky Medical Center ( Site 0561), Tel Aviv
  - Assaf Harofeh Medical Center ( Site 0556), Ẕerifin
- Italy (9):
  - Ospedale San Raffaele-Oncologia Medica ( Site 0309), Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda ( Site 0307), Milan, Lombardy
  - Centro di Riferimento Oncologico CRO ( Site 0304), Aviano, Pordenone
  - Istituto Tumori Giovanni Paolo II ( Site 0306), Bari
  - Policlinico S. Orsola - Malpighi (Bologna) ( Site 0302), Bologna
  - Azienda Ospedaliera per l Emergenza Cannizzaro ( Site 0305), Catania
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 0301), Milan
  - Azienda Ospedaliera Santa Maria ( Site 0303), Terni
  - Ospedale Borgo Roma-Oncologia ( Site 0308), Verona
- Japan (15):
  - Hirosaki University Hospital ( Site 0123), Hirosaki, Aomori
  - National Cancer Center Hospital East ( Site 0128), Kashiwa, Chiba
  - Ehime University Hospital ( Site 0137), Tōon, Ehime
  - Sapporo Medical University Hospital ( Site 0122), Sapporo, Hokkaido
  - University of Tsukuba Hospital ( Site 0126), Tsukuba, Ibaraki
  - Kitasato University Hospital ( Site 0129), Sagamihara, Kanagawa
  - Nara Medical University Hospital ( Site 0133), Kashihara, Nara
  - Saitama Medical University International Medical Center ( Site 0125), Hidaka, Saitama
  - Yamaguchi University Hospital ( Site 0135), Ube, Yamaguchi
  - Akita University Hospital ( Site 0124), Akita
  - Chiba Cancer Center ( Site 0127), Chiba
  - Nagasaki University Hospital ( Site 0136), Nagasaki
  - Osaka City University Hospital ( Site 0132), Osaka
  - Tokushima University Hospital ( Site 0134), Tokushima
  - Medical Hospital, Tokyo Medical And Dental University ( Site 0130), Tokyo
- Netherlands (8):
  - Ziekenhuis Rijnstate ( Site 0342), Arnhem, Gelderland
  - Maastricht Universitair Medisch Centrum - MUMC ( Site 0334), Maastricht, Limburg
  - VieCuri Medisch Centrum ( Site 0340), Venlo, Limburg
  - Amphia Ziekenhuis Breda ( Site 0331), Breda, North Brabant
  - Deventer Ziekenhuis ( Site 0341), Deventer, Overijssel
  - Erasmus MC ( Site 0332), Rotterdam, South Holland
  - Haga Ziekenhuis ( Site 0333), The Hague, South Holland
  - St. Antonius Ziekenhuis ( Site 0335), Utrecht
- Poland (6):
  - Szpital Wojewodzki ( Site 1062), Tarnów, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego ( Site 0535), Wroclaw, Lower Silesian Voivodeship
  - Europejskie Centrum Zdrowia Otwock ( Site 0532), Otwock, Masovian Voivodeship
  - Urologica Praktyka Lekarska Adam Marcheluk ( Site 0543), Siedlce, Masovian Voivodeship
  - Luxmed Onkologia sp. z o. o. ( Site 0541), Warsaw, Masovian Voivodeship
  - Szpital Miejski im. Jana Pawła II w Bielsku-Białej ( Site 0542), Bielsko-Biala, Silesian Voivodeship
- Russia (9):
  - GBUZ Leningrad Regional Clinical Oncology Dispensary ( Site 0426), Kuzmolovskiy Settlement, Leningradskaya Oblast'
  - Russian Scientific Center of Roentgenoradiology ( Site 0424), Moscow, Moscow
  - Central Clinical Hospital with Polyclinic ( Site 0415), Moscow, Moscow
  - Medical Rehabilitation Center ( Site 0411), Moscow, Moscow
  - Murmansk Regional Oncology Dispensary ( Site 0420), Murmansk, Murmansk Oblast
  - Volga District Medical Center Federal Medical and Biological Agency ( Site 0413), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Omsk Clinical Oncology Dispensary ( Site 0418), Omsk, Omsk Oblast
  - Clinical Hospital Saint Luka ( Site 0421), Saint Petersburg, Sankt-Peterburg
  - Yaroslavl Regional SBIH Clinical Oncology Hospital ( Site 0414), Yaroslavl, Yaroslavl Oblast
- South Korea (8):
  - Chonnam National University Hwasun Hospital ( Site 0194), Hwasun Gun, Jeonranamdo
  - National Cancer Center ( Site 0196), Goyang-si, Kyonggi-do
  - Chungnam National University Hospital ( Site 0195), Daejeon, Taejon-Kwangyokshi
  - Korea University Anam Hospital ( Site 0197), Seoul
  - Seoul National University Hospital ( Site 0191), Seoul
  - Severance Hospital ( Site 0192), Seoul
  - Veterans Health Service Medical Center ( Site 0198), Seoul
  - Samsung Medical Center ( Site 0193), Seoul
- Spain (9):
  - Institut Catala d Oncologia Hospital Germans Trias i Pujol ( Site 0351), Badalona, Barcelona
  - ICO L Hospitalet ( Site 0361), L'Hospitalet de Llobregat, Barcelona
  - Xarxa Assistencial Universitaria Manresa ( Site 0354), Manresa, Barcelona
  - Hospital Teresa Herrera - Chuac ( Site 0357), A Coruña, La Coruna
  - Hospital Universitario HM Sanchinarro ( Site 0356), Madrid, Madrid, Comunidad de
  - Hospital Infanta Cristina ( Site 0355), Badajoz
  - Hospital General Universitari Vall d Hebron ( Site 0358), Barcelona
  - Hospital La Princesa ( Site 0862), Madrid
  - Hospital Universitario Gregorio Maranon ( Site 0352), Madrid
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital ( Site 0216), Kaoshiung, Kaohsiung
  - Kaohsiung Chang Gung Memorial Hospital ( Site 0217), Kaohsiung City
  - China Medical University Hospital ( Site 0213), Taichung
  - Taichung Veterans General Hospital ( Site 0214), Taichung
  - National Cheng Kung University Hospital ( Site 0215), Tainan
  - National Taiwan University Hospital ( Site 0211), Taipei
  - Taipei Veterans General Hospital ( Site 0212), Taipei
- Turkey (Türkiye) (8):
  - Cukurova Universitesi Tıp Fakultesi Balcalı Hastanesi ( Site 0457), Adana
  - Ankara Sehir Hastanesi ( Site 0455), Ankara
  - Antalya Memorial Hospital Department of Medical Oncology ( Site 0461), Antalya
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 0454), Istanbul
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 0459), Istanbul
  - Ege Universitesi Tulay Aktas Onkoloji Hastanesi ( Site 0462), Izmir
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi Hastanesi ( Site 0456), Konya
  - Sakarya Universitesi Tip Fakultesi Arastirma Hastanesi ( Site 0460), Sakarya
- United Kingdom (11):
  - Weston Park Hospital ( Site 0387), Sheffield, Derbyshire
  - Queens Hospital-Purple Zone ( Site 0377), Romford, Essex
  - Lister Hospital ( Site 0376), Stevenage, Hertfordshire
  - Kent and Canterbury Hospital ( Site 0390), Canterbury, Kent
  - Royal Preston Hospital ( Site 0379), Preston, Lancashire
  - Saint Bartholomew s Hospital - London ( Site 0386), London, London, City of
  - University College London Hospital NHS Foundation Trust ( Site 0380), London, London, City of
  - Imperial Healthcare NHS Trust Charing Cross Hospital ( Site 0378), London, London, City of
  - Nottingham University Hospital NHS Trust ( Site 0383), Nottingham
  - Derriford Hospital ( Site 0388), Plymouth
  - Royal Stoke University Hospital Univ. Hosps of North Midlands NHST ( Site 0392), Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Matsubara N, de Wit R, Balar AV, Siefker-Radtke AO, Zolnierek J, Csoszi T, Shin SJ, Park SH, Atduev V, Gumus M, Su YL, Karaca SB, Cutuli HJ, Sendur MAN, Shen L, O'Hara K, Okpara CE, Franco S, Moreno BH, Grivas P, Loriot Y. Pembrolizumab with or Without Lenvatinib as First-line Therapy for Patients with Advanced Urothelial Carcinoma (LEAP-011): A Phase 3, Randomized, Double-Blind Trial. Eur Urol. 2024 Mar;85(3):229-238. doi: 10.1016/j.eururo.2023.08.012. Epub 2023 Sep 29. PMID 37778952
- [Derived] Taylor MH, Schmidt EV, Dutcus C, Pinheiro EM, Funahashi Y, Lubiniecki G, Rasco D. The LEAP program: lenvatinib plus pembrolizumab for the treatment of advanced solid tumors. Future Oncol. 2021 Feb;17(6):637-648. doi: 10.2217/fon-2020-0937. Epub 2020 Dec 10. PMID 33300372
- See also: Merck Clinical Trials Information — http://merckclinicaltrials.com/
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26809&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, response/progression or adverse events (AEs) that occurred during the second course of pembrolizumab were not included in efficacy or safety outcome measures.
Groups:
- Pembrolizumab + Lenvatinib: Participants received pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule once daily (QD) until progressive disease (PD) or discontinuation. With protocol amendment 3 (effective: Sep-24-2021), participants discontinued lenvatinib.
  At the investigator's discretion, eligible participants randomized to the pembrolizumab + lenvatinib arm who completed the first course of pembrolizumab or who had stopped pembrolizumab due to confirmed complete response (CR) initiated a second course of pembrolizumab (200 mg IV infusion on Day 1 of each 21-day cycle, for up to 17 cycles [up to approximately 1 additional year]) upon experiencing PD.
- Pembrolizumab + Placebo: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years) PLUS placebo for lenvatinib via oral capsule QD until PD or discontinuation. With protocol amendment 3 (effective: Sep-24-2021), participants discontinued placebo.
  At the investigator's discretion, eligible participants randomized to the pembrolizumab + placebo arm who completed the first course of pembrolizumab, or who had stopped pembrolizumab due to confirmed CR, initiated a second course of pembrolizumab (200 mg IV infusion on Day 1 of each 21-day cycle, for up to 17 cycles [up to approximately 1 additional year]) upon experiencing PD.
Period: Overall Study
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Started | 251 | 254
Treated | 247 | 254
Pembrolizumab + Lenvatinib vs. Pembrolizumab + Placebo Efficacy Analyses | 245 | 242
Pembrolizumab + Lenvatinib vs. Pembrolizumab + Placebo Safety Analyses | 241 | 242
Received Second Course of Pembrolizumab | 2 | 5
Completed | 63 | 77
Not Completed | 188 | 177
Not completed — Death | 178 | 173
Not completed — Physician Decision | 1 | 0
Not completed — Sponsor Decision | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab + Lenvatinib: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule QD until PD or discontinuation. With protocol amendment 3 (effective: Sep-24-2021), participants discontinued lenvatinib.
  At the investigator's discretion, eligible participants randomized to the pembrolizumab + lenvatinib arm who completed the first course of pembrolizumab or who had stopped pembrolizumab due to confirmed CR initiated a second course of pembrolizumab (200 mg IV infusion on Day 1 of each 21-day cycle, for up to 17 cycles [up to approximately 1 additional year]) upon experiencing PD.
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo | Total
Number analyzed (Participants) | 251 | 254 | 505
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.3 (9.3) | 71.9 (8.5) | 72.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 59 | 136
  Male | 174 | 195 | 369
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 10 | 27
  Not Hispanic or Latino | 213 | 218 | 431
  Unknown or Not Reported | 21 | 26 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 78 | 79 | 157
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 164 | 157 | 321
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 9 | 16 | 25
Chemotherapy Ineligibility, Combined Positive Score (CPS), Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — Participants were classified as ineligible for any platinum agent or for cisplatin. CPS=PD-L1 immunohistochemistry positive cell (tumor cell, macrophage, lymphocyte) number divided by total tumor cells expressed as a percentage; classified as CPS ≥10 or <10. ECOG 0=fully active, ECOG 1=strenuous activity restricted, ECOG 2=in bed <50% of time; classified as ECOG=2 or 0/1. Per protocol stratification: (1) Ineligible for any platinum agents CPS ≥10 ECOG 2; (2) Ineligible for any platinum agents CPS <10 ECOG 2; (3) Cisplatin-ineligible CPS ≥10 ECOG 2; (4) Cisplatin-ineligible CPS ≥10 ECOG 0 or 1.
  Participants
    Ineligible for any platinum agents CPS ≥10 ECOG 2 | 83 | 84 | 167
    Ineligible for any platinum agents CPS <10 ECOG 2 | 118 | 120 | 238
    Cisplatin-ineligible CPS ≥10 ECOG 2 | 8 | 8 | 16
    Cisplatin-ineligible CPS ≥10 ECOG 0 or 1 | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to the first documented PD per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) by blinded independent central review (BICR), or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS as assessed by BICR per RECIST 1.1 is presented. Protocol-specified final analysis for this primary outcome measure was performed with an analysis data cut-off date of Jul-26-2021.
Time Frame: Up to approximately 25 months
Population: All participants randomized prior to the protocol-specified primary completion analysis data cut-off.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab + Lenvatinib: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule QD until PD or discontinuation. With protocol amendment 3 (effective: Sep-24-2021), participants discontinued lenvatinib.
  At the investigator's discretion, eligible participants randomized to the pembrolizumab PLUS lenvatinib arm who completed the first course of pembrolizumab or who had stopped pembrolizumab due to confirmed CR initiated a second course of pembrolizumab (200 mg IV infusion on Day 1 of each 21-day cycle, for up to 17 cycles [up to approximately 1 additional year]) upon experiencing PD.
- Pembrolizumab + Placebo: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years) PLUS placebo for lenvatinib via oral capsule QD until PD or discontinuation. With protocol amendment 3 (effective: Sep-24-2021), participants discontinued placebo.
  At the investigator's discretion, eligible participants randomized to the pembrolizumab PLUS placebo arm who completed the first course of pembrolizumab or who had stopped pembrolizumab due to confirmed CR initiated a second course of pembrolizumab (200 mg IV infusion on Day 1 of each 21-day cycle, for up to 17 cycles [up to approximately 1 additional year]) upon experiencing PD.
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 245 | 242
Months | 4.5 [4.0 to 6.0] | 4.0 [2.7 to 5.4]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Superiority; p = 0.4107, Log Rank — Two-sided p-value based on log rank test stratified on chemotherapy ineligibility, programmed cell death ligand 1 (PD-L1) CPS, and ECOG performance status (PS); Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.72 to 1.14] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified on chemotherapy ineligibility, PD-L1 CPS, and ECOG PS

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were to be censored at the date of the last follow-up. Protocol-specified final analysis for this primary outcome measure was performed with an analysis data cut-off date of Jul-26-2021.
Time Frame: Up to approximately 25 months
Population: All participants randomized prior to the protocol-specified primary completion analysis data cut-off.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 245 | 242
Months | 11.8 [9.1 to 15.1] | 12.9 [9.8 to 17.8]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Superiority; p = 0.3505, Log Rank — Two-sided p-value based on log rank test stratified on chemotherapy ineligibility, PD-L1 CPS, and ECOG PS; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.87 to 1.48] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a confirmed CR (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by BICR. The percentage of participants who experienced a CR or PR is presented. Protocol-specified final analysis for this secondary outcome measure was performed with an analysis data cut-off date of Jul-26-2021.
Time Frame: Up to approximately 25 months
Population: All participants randomized prior to the protocol-specified primary completion analysis data cut-off.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 245 | 242
Percentage of Participants | 33.1 [27.2 to 39.3] | 28.9 [23.3 to 35.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Superiority; Difference in Percentage = 4.1, 95% CI 2-sided [-4.0 to 12.2] — Based on Miettinen & Nurminen method stratified on chemotherapy ineligibility, PD-L1 CPS, and ECOG PS

4. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrated a confirmed CR (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by BICR, DOR was defined as the time from first documented evidence of a CR or PR until PD or death. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions as well as an absolute increase of ≥5 mm in the sum of diameters. The appearance of one or more new lesions was also considered PD. The DOR as assessed by BICR per RECIST 1.1 for participants who experienced a confirmed CR or PR is presented. Protocol-specified final analysis for this secondary outcome measure was performed with an analysis data cut-off date of Jul-26-2021.
Time Frame: Up to approximately 25 months
Population: All participants randomized prior to the protocol-specified primary completion analysis data cut-off and who also experienced a confirmed CR or partial response.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 81 | 70
Months | NA [NA to NA] — NA = Median, upper limit and lower limit of range could not be reached at time of data cut-off due to insufficient number of responding participants with relapse. | NA [NA to NA] — NA = Median, upper limit and lower limit of range could not be reached at time of data cut-off due to insufficient number of responding participants with relapse.

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who have a CR (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) or stable disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD [PD: ≥20% increase in the sum of diameters of target lesions and an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD]). DCR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. The DCR as assessed by BICR per RECIST 1.1 is presented. Protocol-specified final analysis for this secondary outcome measure was performed with an analysis data cut-off date of Jul-26-2021.
Time Frame: Up to approximately 25 months
Population: All participants randomized prior to the protocol-specified primary completion analysis data cut-off.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 245 | 242
Percentage of Participants | 66.9 [60.7 to 72.8] | 56.2 [49.7 to 62.5]

6. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (GHS) (Item 29) and Quality of Life (QOL) (Item 30) Combined Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions regarding GHS ("How would you rate your overall health during the past week?") and QOL ("How would you rate your overall quality of life during the past week?") were scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores were standardized, so that scores range from 0 to 100. The change from baseline in GHS (EORTC QLQ-C30 Item 29) and QOL (EORTC QLQ-C30 Item 30) combined score is presented. A higher score indicates a better outcome. Final analysis for this secondary outcome measure was performed with an analysis data cut-off date of Jul-26-2021, as specified in the Supplemental Statistical Analysis Plan (sSAP).
Time Frame: Baseline and Week 11
Population: All participants who were randomized and received at least one dose of study treatment prior to the primary completion analysis data cut-off and who also had data available from at least 1 EORTC QLQ-C30 Item 29 and 30 assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 240 | 231
Scores on a scale | 0.73 [-2.63 to 4.09] | 3.79 [0.47 to 7.12]
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other; p = 0.182, cLDA model — Two-sided p-value based on log rank test stratified on chemotherapy ineligibility, PD-L1 CPS, and ECOG PS; Difference in least squares means = -3.07, 95% CI 2-sided [-7.57 to 1.44] — Based on a constrained longitudinal data analysis (cLDA) model with the PRO scores as the response variable with covariates for treatment by study visit interaction, and stratification factors by chemotherapy ineligibility, PD-L1 CPS, and ECOG PS

7. Secondary Outcome: Time to True Deterioration (TTD) Based on Change From Baseline in EORTC QLQ-C30 GHS (Item 29) and QOL (Item 30) Combined Score
Description: TTD was defined as the time from baseline to the first onset of a ≥10-point negative change (decrease) from baseline in GHS (EORTC QLQ-C30 Item 29) & QOL (EORTC QLQ-C30 Item 30) combined score. The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions regarding GHS ("How would you rate your overall health during the past week?") and QOL ("How would you rate your overall quality of life during the past week?") were scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores were standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from baseline in GHS and QOL combined score, is presented. A longer TTD indicates a better outcome. Final analysis for this secondary outcome measure was performed with an analysis data cut-off date of Jul-26-2021, as specified in the sSAP.
Time Frame: Baseline and up to approximately 25 months
Population: All participants who were randomized and received at least one dose of study treatment prior to the primary completion analysis data cut-off and who also had data available from baseline and ≥1 post-baseline EORTC QLQ-C30 Item 29 and 30 assessments.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 233 | 226
Months | 3.4 [2.1 to 4.3] | 7.6 [4.2 to NA] — NA = Upper limit was not reached at time of data cut-off due to an insufficient number of participants having the first onset of a ≥10-point negative change (decrease) from baseline in GHS (EORTC QLQ-C30 Item 29) & QOL (EORTC QLQ-C30 Item 30) combined score.
Statistical Analysis 1: Comparison: Pembrolizumab + Lenvatinib vs Pembrolizumab + Placebo; Test type: Other; p = 0.0005, Log Rank — Two-sided p-value based on log rank test stratified on chemotherapy ineligibility, PD-L1 CPS, and ECOG PS; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [1.24 to 2.16] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by chemotherapy ineligibility, PD-L1 CPS, and ECOG PS

8. Secondary Outcome: Number of Participants Who Experience an AE
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE is presented. Final analysis for this secondary outcome measure was performed with an analysis data cut-off date of Jul-26-2021.
Time Frame: Up to approximately 25 months
Population: All participants who were randomized and received at least one dose of study treatment prior to the primary completion analysis data cut-off.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 241 | 242
Participants | 234 | 235

9. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study treatment due to an AE is presented. Final analysis for this secondary outcome measure was performed with an analysis data cut-off date of Jul-26-2021.
Time Frame: Up to approximately 25 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Lenvatinib | Pembrolizumab + Placebo
Number analyzed (Participants) | 241 | 242
Participants | 83 | 44

ADVERSE EVENTS:
Time Frame: Up to approximately 52 months
Description: All-Cause Mortality (ACM) includes all randomized participants. AEs include all randomized participants who received ≥1 dose of study treatment. Progression of the cancer under study was not considered an AE unless related to study drug. MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs. Data are reported by treatment received. ACM and AEs are reported separately for pembrolizumab second course.
Groups:
- Lenvatinib + Pembrolizumab First Course: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years) PLUS lenvatinib 20 mg via oral capsule QD until PD or discontinuation. With protocol amendment 3 (effective: Sep-24-2021), participants discontinued lenvatinib.
- Placebo + Pembrolizumab First Course: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 21-day cycle for up to 35 cycles (up to approximately 2 years) PLUS placebo for lenvatinib via oral capsule QD until PD or discontinuation.
  With protocol amendment 3 (effective: Sep-24-2021), participants discontinued placebo.
- Lenvatinib + Pembrolizumab → Pembrolizumab Second Course: At the investigator's discretion, eligible participants randomized to the pembrolizumab PLUS lenvatinib arm who completed the first course of pembrolizumab, or who had stopped pembrolizumab due to confirmed CR, initiated a second course of pembrolizumab (200 mg IV infusion on Day 1 of each 21-day cycle, for up to 17 cycles [up to approximately 1 additional year]) upon experiencing PD.
- Placebo + Pembrolizumab → Pembrolizumab Second Course: At the investigator's discretion, eligible participants randomized to the pembrolizumab PLUS placebo arm who completed the first course of pembrolizumab, or who had stopped pembrolizumab due to confirmed CR, initiated a second course of pembrolizumab (200 mg IV infusion on Day 1 of each 21-day cycle, for up to 17 cycles [up to approximately 1 additional year]) upon experiencing PD.
Arm/Group | Lenvatinib + Pembrolizumab First Course | Placebo + Pembrolizumab First Course | Lenvatinib + Pembrolizumab → Pembrolizumab Second Course | Placebo + Pembrolizumab → Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 178/251 | 175/254 | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 155/247 | 116/254 | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 238/247 | 236/254 | 1/2 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab First Course (N=247) | Placebo + Pembrolizumab First Course (N=254) | Lenvatinib + Pembrolizumab → Pembrolizumab Second Course (N=2) | Placebo + Pembrolizumab → Pembrolizumab Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 7 (7) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 14 (14) | 5 (5) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 4 (5) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 9 (9) | 14 (17) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 4 (6) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular access site occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic enzymes increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 2 (3) | 3 (3) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lead dislodgement (Product Issues) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 12 (17) | 5 (5) | 0 (0) | 0 (0)
Bladder mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 6 (7) | 5 (5) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perinephric collection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenvatinib + Pembrolizumab First Course (N=247) | Placebo + Pembrolizumab First Course (N=254) | Lenvatinib + Pembrolizumab → Pembrolizumab Second Course (N=2) | Placebo + Pembrolizumab → Pembrolizumab Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 48 (57) | 64 (74) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 16 (17) | 12 (13) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 98 (109) | 27 (30) | 0 (0) | 0 (0)
Xerophthalmia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 25 (32) | 23 (26) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 14 (17) | 11 (12) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 40 (50) | 38 (45) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 65 (111) | 51 (75) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 52 (65) | 44 (53) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 18 (23) | 7 (10) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 37 (42) | 26 (31) | 0 (0) | 1 (1)
Asthenia (General disorders) | 52 (62) | 33 (46) | 0 (0) | 0 (0)
Fatigue (General disorders) | 52 (58) | 53 (55) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 20 (21) | 9 (9) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 28 (31) | 26 (27) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 25 (33) | 35 (47) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 3 (3) | 8 (9) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 7 (10) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 54 (75) | 46 (66) | 0 (0) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 22 (29) | 15 (19) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 24 (33) | 27 (39) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 21 (25) | 17 (20) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 19 (21) | 16 (16) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 4 (5) | 11 (16) | 0 (0) | 2 (5)
Blood creatinine increased (Investigations) | 28 (33) | 19 (27) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 39 (49) | 28 (40) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 16 (23) | 7 (10) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 50 (51) | 23 (24) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 68 (85) | 43 (51) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (12) | 12 (15) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (12) | 16 (18) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 19 (22) | 12 (12) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 18 (21) | 17 (19) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (38) | 26 (31) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (27) | 21 (24) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (14) | 4 (4) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (15) | 10 (10) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 21 (25) | 14 (16) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 12 (12) | 17 (18) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 3 (3) | 6 (9) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 32 (36) | 32 (47) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 101 (149) | 71 (94) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 14 (22) | 9 (11) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 20 (26) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 40 (49) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 15 (20) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 25 (29) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 34 (41) | 48 (64) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 38 (52) | 27 (33) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 99 (125) | 23 (33) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 10 (12) | 13 (15) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT03898180/Prot_001.pdf
  • Statistical Analysis Plan (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT03898180/SAP_002.pdf